CLINICAL TRIAL: NCT06478290
Title: Pilot Assessment of the Safety of a Combination of Curcumin, Omega-3, and Vitamin D Supplements (PASCOD) in ACPA+ Individuals
Brief Title: Pilot Assessment of the Safety of a Combination of Curcumin, Omega-3, and Vitamin D Supplements in ACPA+ Individuals
Acronym: PASCOD3
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HS26482 (B2024:059)
Record Dates: First submitted 2024-06-13; First posted 2024-06-27 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Healthy Participants
Keywords: Rheumatoid Arthritis; Curcumin; Omega-3; Vitamin D
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Curcumin; Docosahexaenoic Acids; Vitamin D

STUDY DESIGN:
Intervention Model Description: This pilot study will have an open label pre-post design, so no randomization or blinding of treatment (COD) will occur.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Theracurmin, Vitamin D, and Omega-3 (Experimental): Theracurmin Double Strength: 180 mg/day (oral, 3 tablets of 60 mg taken by mouth) Vitamin D: 2000 IU/day LipoMicel (oral, 1 tablet taken by mouth) Omega-3: 900 mg day (oral, 1 tablet taken by mouth)
  Interventions: Combination Product: curcumin, omega-3, and vitamin D (COD)

INTERVENTIONS:
Combination Product: curcumin, omega-3, and vitamin D (COD) — Combination of curcumin, omega-3, and vitamin D supplements (COD). Theracurmin Double Strength/Natural Factors Canada 180 mg/day (oral, 3 tablets of 60 mg taken by mouth) Vitamin D: 2000 IU/day LipoMicel/Natural Factors Canada (oral, 1 tablet taken by mouth) Omega-3: 900 mg day (oral, 1 tablet taken by mouth)

SUMMARY:
The goal of this clinical trial is to determine if the level of Anti-cyclic citrullinated peptide antibody (ACPA) is altered after taking curcumin, omega-3, and vitamin D supplements (COD) for 3 months. It will also determine the safety and tolerability of COD in the study population. This trial aims to answer the following questions: Does COD consumption lower the level of ACPA in the study participants? What side effects will participants have after taking COD? This pilot study will have an open label pre-post design and study participants will know that they are using each of the three supplements. Participants will: Take the combination of supplements following an evening meal, for 84 consecutive days. Visit the clinic/study team twice during the study duration on days 0 and 84 for checkups and tests. Keep a diary of study treatment consumption.

DETAILED DESCRIPTION:
Rheumatoid Arthritis (RA) is a prevalent autoimmune disease. Curcumin formulations are recognized for their potent anti-inflammatory effects, mainly targeting NF-kB signaling. Supplementation with Acumin™ has shown significant benefits for RA patients, including pain relief, reduced morning stiffness, and improved joint function, alongside decreases in inflammatory markers and autoantibody levels. In murine arthritis models, a bioavailable curcumin form, combined with a diet rich in vitamin D and omega-3, notably altered disease progression. Therefore, a pilot trial is set for anti-cyclic citrullinated peptide antibody+ (APCA+) individuals without RA. The primary objective of this study will determine if the level of ACPA is altered after taking curcumin, omega-3, and vitamin D (COD) for 3 months. The secondary objective is to determine the safety and tolerability of COD in the study population. Exploratory outcomes will include assessment of joint, symptoms, blood biochemistry and hematology. This study will enroll 50 ACPA+ individuals without RA, aiming for an equal distribution of male and female participants. Participants identified as ACPA+ from the RA Auto-antibody Detection study (RAAD) will undergo eligibility screening. The study will involve open-label administration of ACUMIN™ Turmeric Complex (500 mg), Omega-3 (900 mg), and Vitamin D3 (2500 IU) once daily for 84 consecutive days. Joint examinations will be conducted by a study physician, and blood specimens will be collected by certified phlebotomists at designated sites. Trained personnel will handle questionnaire surveys, anthropometrics, follow-ups, and coordinating visits. Data will be recorded on paper-based CRFs and entered into the secure REDCap database. The trial will take place at Health Sciences Centre (MS7) in Winnipeg for urban participants and in First Nation communities with established research agreements with the team (Norway House First Nation).

ELIGIBILITY:
Inclusion Criteria

* Verified to be ACPA+ based on serum testing
* Age 18 to 65 years old
* Willing to provide contact information by email, telephone and mailing address
* Participant agrees to take the supplements every day for 84 days
* Female participants of child-bearing potential must be willing to ensure that they use contraception during the trial
* Participant has clinically acceptable laboratory results including routine hematology (CBC) and biochemistry (electrolytes, creatinine, ALT, ALP, GGT, AST, Glucose)
* In the Investigator's opinion, is able and willing to comply with all trial requirements
* If participant is currently taking curcumin, vitamin D and/or omega-3 supplements they must agree to a washout period of at least 1 month prior to the start of the trial.
* Participant agrees to be followed longitudinally in the PRE-RA cohort study, following the completion of this trial.
* Participant is willing and able to give free informed consent and written consent in English, for participation in the trial.

Exclusion Criteria

The participant may not enter the trial if ANY of the following apply:

* Current use of warfarin or similar anticoagulant medication (at the discretion of the P.I.)
* Female participant who is pregnant, lactating or planning pregnancy during the course of the trial
* Female of childbearing potential who is unwilling to use contraception during the trial
* Scheduled elective surgery or other procedures requiring general anaesthesia during the trial
* Any significant disease or disorder which, in the opinion of the Investigator, may either put the participant at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.
* Concurrent commitment to enroll in another clinical trial
* Regular consumption of vitamin D, omega-3, curcumin supplements and/or curcumin containing product within the last 3 months and unwilling to stop consumption for at least a month prior to the start of the trial.
* Self-report of allergic reaction to fish
* Participants who indicate that they will not consume the treatments on a daily basis
* Current consumption of > 14 drinks per week, (1 drink = 12oz of beer, 5oz of wine or 1.5oz distilled spirits)
* Participants who report they have had viral or bacterial infection in the last 4 weeks (e.g. COVID-19, the flu, a cold, stomach flu, bladder infection, strep throat), and are not fully recovered. Once fully recovered they can participate.
* Participant has been recently vaccinated (past 4 weeks). Participant can continue in the trial 1-month after receiving the vaccination.
* Has vacation/s planned during the trial that may interfere with study monitoring and visit 2. The start of the trial can be adjusted to accommodate planned vacations.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
ACPA levels | At Day 0 and Day 84
  Anti-cyclic citrullinated peptide antibody (ACPA) levels will be determined with a CCP3.1 ELISA

SECONDARY OUTCOMES:
Side-effect profile of COD | At Day 0 and Day 84
  Side-effect profile and prevalence of side-effects of Theracurmin Double Strength, Omega-3, and Vitamin D supplementation will be determined through monitoring the blood results for biochemical and haematology analysis

OTHER OUTCOMES:
Waist circumference measures | At Day 0 and Day 84
  Waist circumference in cm using a measuring tape
Weight measures | At Day 0 and Day 84
  Weight in kg using a scale
Height measures | At Day 0 and Day 84
  Height in cm using a measuring tape
Blood pressure measures | At Day 0 and Day 84
  Systolic and diastolic Blood pressure will be measured in mmHg using blood pressure machine
Tender and Swollen Joint Counts (TSJC) | At Day 0 and Day 84
  44 tender and swollen joint count will be performed by a rheumatologist
SDAI | At Day 0 and Day 84
  Simple Disease Activity Index (SDAI) assessment will be used to determine severity of RA using clinical and laboratory data
CDAI | At Day 0 and Day 84
  Clinical Disease Activity Index (CDAI) assessment will be used to determine severity of RA using clinical and laboratory data
DAS28-CRP | At Day 0 and Day 84
  The Disease Activity Score (DAS28)-CRP will be determined to assess RA disease activity, calculated once the C-reactive protein (CRP) result is available
Hand grip strength | At Day 0 and Day 84
  Hand grip strength will be measured using a Dynamometer in kg, taken in triplicate
RAPID3 | At Day 0 and Day 84
  Routine assessment of patient index data. Disease activity index calculated from a short and questionnaire
White blood cells (WBC) | At Day 0 and Day 84
  WBC measured in x10^9/L
Hemoglobin | At Day 0 and Day 84
  Hemoglobin measured in g/L
Platelets | At Day 0 and Day 84
  Platelets measured in x10^9/L
Mean platelet volume (MVP) | At Day 0 and Day 84
  MVP measured in fL
BUN | At Day 0 and Day 84
  The total blood urea concentration in mmol/L
Magnesium | At Day 0 and Day 84
  Magnesium measured in mmol/L
Lipid profile | At Day 0 and Day 84
  Total cholesterol, LDL, HDL, and Non-fasted triglycerides will be measured in mmol/L
Albumin | At Day 0 and Day 84
  Total blood albumin concentration in g/L
Total and direct bilirubin | At Day 0 and Day 84
  Total and direct bilirubin is measured in μmol/L
Sodium | At Day 0 and Day 84
  Total blood sodium concentration in mmol/L
Potassium | At Day 0 and Day 84
  Total blood potassium concentration in mmol/L
Chloride | At Day 0 and Day 84
  Total blood chloride concentration in mmol/L
Bicarbonate HCO3 | At Day 0 and Day 84
  Bicarbonate measured in mmol/L
Creatinine | At Day 0 and Day 84
  Total blood creatinine concentration in μmol/L
AST | At Day 0 and Day 84
  AST is measured in U/L
ALT | At Day 0 and Day 84
  ALT is measured in U/L
ALP | At Day 0 and Day 84
  ALP is measured in U/L
GGT | At Day 0 and Day 84
  GGT is measured in U/L
Glucose | At Day 0 and Day 84
  Total fasted blood glucose concentration in mmol/L
Calcium | At Day 0 and Day 84
  Total blood calcium concentration in mmol/L
Phosphate (PO4) | At Day 0 and Day 84
  Total blood phosphate concentration in mmol/L
CRP | At Day 0 and Day 84
  C-Reactive Protein (CRP)

CONTACTS AND LOCATIONS:
Overall Officials: Liam O'Neil, MD, MHSc, Principal Investigator — University of Manitoba
Locations (2):
- Canada (2):
  - Norway House Health Centre, Norway House, Manitoba
  - Health Sciences Centre, Winnipeg, Manitoba

IPD SHARING:
Plan to Share IPD: Undecided